CLINICAL TRIAL: NCT04973059
Title: Determining Levels of Enhanced Function Associated With the Permobil SmartDrive Manual Wheelchair Power Assist
Brief Title: Determining Levels of Function Associated With Permobil SmartDrive Manual Wheelchair Assist
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Permobil, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Pro00106859
Record Dates: First submitted 2021-06-16; First posted 2021-07-22 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-10

CONDITIONS: Wheelchairs
Keywords: wheelchair; participation; accessibility; power assist; overuse injury
MeSH Terms: conditions — Cumulative Trauma Disorders

STUDY DESIGN:
Intervention Model Description: This study is not evaluating a clinical intervention. There is no anticipated clinical benefit from this study. It is assessing whether use of the SmartDrive increases participation and decreases solution isolation. Secondarily it is will provide information about the levels of exertion needed in comparing wheelchair propulsion using SmartDrive and usual wheelchair propulsion. We intend to determine if SmartDrive improves participation in the winter when it is difficult to propel manual wheelchair on snow covered sidewalks and parking lots. Participants will be randomly assigned to using either the SmartDrive or not in the first week of monitoring in the summer. They will then switch to either the intervention (SmartDrive) or control (no SmarDrive) for the next week. This will then be repeated in the winter. Activity information will be collected using the SmartDrive sensor and another sensor that will measure a wide range of activity data including for the control arm of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Summer Conditions with SmartDrive (Active Comparator): This arm is with the participant using the SmartDrive during a week in the summer. The SmartDrive is a manual wheelchair accessory that provide power assistance to reduce the necessary level of propulsion force. The goal is to increase participation by reducing propulsion effort.
  Interventions: Device: SmartDrive Summer
- Summer Conditions activity measurement only (No Intervention): This arm is with the participant using their wheelchair during a week in the summer no power assist.
- Winter Conditions activity measurement only (No Intervention): This arm is with the participant using their wheelchair during a week in the winter no power assist
- Winter Conditions with SmartDrive (Active Comparator): This arm is with the participant using the SmartDrive during a week in the winter. The SmartDrive is a manual wheelchair accessory that provide power assistance to reduce the necessary level of propulsion force. The goal is to increase participation by reducing propulsion effort.
  Interventions: Device: SmartDrive Winter

INTERVENTIONS:
Device: SmartDrive Summer — The SmartDrive is a power assist accessory for a manual wheelchair
  Arms: Summer Conditions with SmartDrive
Device: SmartDrive Winter — The SmartDrive is a power assist accessory for a manual wheelchair
  Arms: Winter Conditions with SmartDrive

SUMMARY:
This study will determine whether a power assist accessory for manual wheelchairs increases participation in community activities. This study will determine whether the power assist device (SmartDrive) is effective by increase participating in both winter and summer conditions.

DETAILED DESCRIPTION:
The University of Alberta, Faculty of Rehabilitation Medicine Rehabilitation Robotics Laboratory undertakes a wide range of research relating to wheelchair propulsion. They have developed a sensor (Redliner ) that measures levels of exertion associated with wheelchair ambulation during everyday activities. The device is linked to the user's cell phone and records a wide range of clinically relevant parameters continuously linking them to the GPS (global positioning system) coordinates of the wheelchair user. This device has significant advantages over more sophisticated wheelchair propulsion force measuring devices such as SmartWheel which are heavy and intended for clinic-based measurements. Redliner fits onto the wheels of any manual wheelchair and its low cost lends itself to clinical studies that are fully powered statistically.

Permobil have developed a product, SmartDrive, that can be retrofitted to a manual wheelchair to provide assistance in propelling the wheelchair. It is paired to PushTracker E2 which communicates with the SmartDrive to record parameters such as location, distance travelled, speed and provides a convenient way to control the SmartDrive which is located between the rear wheels of the wheelchair.

The cost of the SmartDrive at US$6,500 exceeds that of most publicly funded manual wheelchairs but is much less than most powered wheelchairs. For manual wheelchair users the SmartDrive is intended to reduce the risk of upper extremity overuse injuries and enables wheelchair users who are marginally functional for community ambulation to achieve their goals, without substantial investment and the collateral costs of transportation and home modifications that a powered wheelchair entails.

One of the challenges of the SmartDrive technology is that the data that has been collected so far is not benchmarked against the performance of wheelchair users prior to acquiring the power assist capability. The "value added" by the device to the user is therefore primarily anecdotal. With the objective of ensuring this technology is widely available, including through public and employer funded benefits, criteria to indicate the level of benefit achieved with SmartDrive are needed. These in turn could be translated into eligibility criteria to be used by both wheelchair users and funders. Redliner could then be used routinely to collect baseline data for wheelchair users wishing to obtain a SmartDrive to determine this eligibility.

This study will compare the benefits of the SmartDrive in the challenging winter conditions in Edmonton and then in the Spring when snow cover has melted. Many wheelchair users in Canada report social isolation due to winter conditions, particularly associated with snow covered sidewalks and streets and this study could demonstrate a particular benefit of the SmartDrive.

The proposed project will bring together our Redliner technology with the SmartDrive/Pushtracker E2 in a complimentary manner in a carefully designed clinical trial of active manual wheelchair users. The study design will be a longitudinal (1 week), repeated measures, cohort, intervention cross-over trial conducted in winter and non-winter conditions. The order of the intervention (SmartDrive use) will be randomized. Both the SmartDrive and Redliner will provide measures of community functioning.

ELIGIBILITY:
Inclusion Criteria:

* Active wheelchair user using a wheelchair as their primary means of mobility (at least 4 hours each day)
* Capable of giving signed informed consent which includes compliance with the requirements listed in the informed consent form (ICF) and in this protocol
* 18 years of age inclusive, at the time of signing the informed consent.
* If the participant has a spinal cord injury Motor level C6-L3 Spinal Cord Injury, American Spinal Injury Association Impairment Scale (AIS) A-C since at least six months
* Full time manual wheelchair users, able to propel their own wheelchairs independently
* Eligible reason for SmartDrive prescription (Self-reported shoulder pain, and/or decreased physical endurance for propulsion, limiting user from activity)

Exclusion Criteria:

* Uncontrolled exercise-induced asthma
* Heart condition or high blood pressure
* Chest pain at rest, during physical activity, or during physical activity
* Severe visual impairment that requires an attendant or guide dog
* Cognitive impairment affecting the ability to operate the SmartDrive, indicated by participant's clinician
* Weigh more than 150 Kg due to the technical specification of the SmartDrive
* Currently participating in another clinical study anticipated to affect the outcome or ability to compete this study
* Planned change from daily routines during the measurement periods, such as holiday, move, change jobs
* For any other reason not suitable for participation in the study indicated by participant's clinician
* Do not use a smart phone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-09-04 (Actual)

PRIMARY OUTCOMES:
Wheelchair User's Shoulder Pain Index (WUSPI) change is being assessed | Arm 1: Applied after 7 days of Use. Arm 2: Applied after 7 days of Use. Arm 3: Applied after 7 days of Use. Arm 4: Applied after 7 days of Use.
  Wheelchair Users' Pain Index Range 0 - 150 VAS high values indicate higher pain

OTHER OUTCOMES:
Wheelchair Users Outcome Measure (WhOM) change is being assessed | Arm 1: Applied after 7 days of Use. Arm 2: Applied after 7 days of Use. Arm 3: Applied after 7 days of Use. Arm 4: Applied after 7 days of Use.
  Wheelchair Users Outcome Measure Range 0-100 high values indicate high level of satisfaction with wheelchair participation/activity

CONTACTS AND LOCATIONS:
Overall Officials: Martin Ferguson-Pell, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Hopkins JE, Selby ET, Shandal RK, Martin N, Ferguson-Pell M, Armstrong E. The effects of the SmartDrive on fostering participatory opportunities for manual wheelchair users: a qualitative exploration. Disabil Rehabil Assist Technol. 2025 Oct;20(7):2500-2509. doi: 10.1080/17483107.2025.2488387. Epub 2025 Apr 8. PMID 40197107